CLINICAL TRIAL: NCT07118423
Title: Effects of Resistance Training in Centenarians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Collaborators: University of Castilla-La Mancha (Other)
Responsible Party: Principal Investigator, Adrián Hernández-Vicente, PhD, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #PI18/381
Record Dates: First submitted 2025-07-14; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Frailty; Muscle Power; Old and Very Old People; Cognitive Abilities; Physical Activity
MeSH Terms: conditions — Frailty; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): The exercise group performed twice per week, nonconsecutive, resistance training over 12 weeks. Exercise sessions consisted of 1-3 sets of the 8-exercise routine at 50-70% of the estimated one-repetition maximum.
  Interventions: Other: Exercise
- Control group (No Intervention): The control group received the usual care in nursing homes.

INTERVENTIONS:
Other: Exercise — The intervention group performed twice per week, nonconsecutive, resistance training over 12 weeks. The sessions consisted of 1-3 sets of eight exercises at 50-70% of the estimated one-repetition maximum.
  Arms: Exercise group

SUMMARY:
This study is a multicenter intervention evaluating the effectiveness and safety of resistance training in institutionalized centenarians.

The aim of the study is to analyze the effects of 12 weeks of resistance training on frailty, muscle power, physical function, strength, functional independence, physical activity, cardiovascular health, cognitive function, and quality of life in adults aged 100 and over living in nursing homes.

DETAILED DESCRIPTION:
Although exercise interventions have shown benefits in octogenarians and nonagenarians, their potential for improving predictors of healthy ageing has not yet been explored in institutionalized centenarians

The aim of the study is to analyze the effects of 12 weeks of resistance training on frailty, muscle power, physical function, strength, functional independence, physical activity, cardiovascular health, cognitive function, and quality of life in adults aged 100 and over living in nursing homes.

ELIGIBILITY:
Inclusion Criteria:

* Women and men aged 100 years and over living in geriatric nursing homes.

Exclusion Criteria:

* Participants were excluded if they were bedridden, going through an acute disease or presented any clinical condition contraindicating physical exercise as outlined in the American College of Sports Medicine's Guidelines.

Min Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Frailty using Fried's Frailty Criteria | T0 (baseline) and T1 (post 12 weeks)
  Fried's frailty phenotype is based on five criteria (habitual gait speed, handgrip strength , involuntary weight loss, exhaustion and low physical activity). The score ranges from 0 to 5, where each criterion met counts as one point. A score of 0 indicates best status, while a score of 5 indicates worst status.
Frailty using Frailty Trait Scale - Short Form | T0 (baseline) and T1 (post 12 weeks)
  Frailty Trait Scale - Short Form evaluates 5 domains, including body mass index, physical activity, static balance, habitual gait speed and handgrip strength. The score ranges from 0 to 50, where each criterion met counts as one point. A score of 0 indicates best status, while a score of 50 indicates worst status.
Muscle power | T0 (baseline) and T1 (post 12 weeks)
  Muscle power assessed in 30-s sit-to-stand test.
Physical function based on the Short Physical Performance Battery | T0 (baseline) and T1 (post 12 weeks)
  The Short Physical Performance Battery is based on the ability to stand with the feet together in the side-by-side, semi-tandem, and tandem positions, time to walk 4 meters, and time to rise from a chair and return to the seated position 5 times. The score ranges from 0 to 12 points. Higher scores indicate better physical function, while lower scores reflect poorer physical function.
Physical function using Physical Performance Mobility Examination. | T0 (baseline) and T1 (post 12 weeks)
  The Physical Performance Mobility Examination includes six mobility tasks integral to daily life: bed mobility, transfer skills, multiple stands from chair, standing balance, step-up, and ambulation. The score ranges from 0 to 12 points. Higher scores indicate better physical function, while lower scores reflect poorer physical function.
Physical function based on the gait speed in 6 meters. | T0 (baseline) and T1 (post 12 weeks)
  Gait speed is measured in meters per second (m/s). Higher values indicate better mobility.
Physical function using the Time Up and Go test. | T0 (baseline) and T1 (post 12 weeks)
  The Timed Up and Go test measures the time it takes participants to stand up, walk 3 meters, turn around, and sit back down. Shorter times reflect better mobility
Cognitive function using Mini Mental State Examination. | T0 (baseline) and T1 (post 12 weeks)
  Mini Mental State Examination questionnaire incorporates 11 items that measure attention and orientation, memory, registration, recall, calculation, language, and ability to draw a complex polygon, and results in scores ranging from 1 (lowest cognitive function) to 30 (highest cognitive function) points.
Cognitive function using the animal naming test within 1 minute. | T0 (baseline) and T1 (post 12 weeks)
  In the animal naming test, participants are asked to name as many animals as possible in 60 seconds. The higher number of correctly named reflects better cognitive function.
Cognitive function using the clock drawing test. | T0 (baseline) and T1 (post 12 weeks)
  The score in the clock drawing test ranges from 0 to 10. This score evalutes visuospatial skills, executive functions, and the ability to follow instructions. Higher scores indicate better cognitive function.
Quality of life using EuroQoL-5 Dimension questionnaire. | T0 (baseline) and T1 (post 12 weeks)
  EuroQoL-5D Index ranges from a value of 1 (best state of health) to 0 (death). Although there are negative values for the index, corresponding to those states of health that are valued as worse than death.
Quality of life using Visual Analog Scale. | T0 (baseline) and T1 (post 12 weeks)
  Visual Analog Scale evaluates self-reported quality of life on a vertical scale ranging from 0 (worst health) to 100 (best health). This score provides a subjective measure of the patient's perception of their current health status.
Isometric muscle strength | T0 (baseline) and T1 (post 12 weeks)
  Maximum voluntary isometric strength in handgrip, knee extension, elbow flexion and should abduction, measured using a dynamometer.
Disability | T0 (baseline) and T1 (post 12 weeks)
  The Barthel index is a 10-item questionnaire that provides information about the autonomy to cook food, wash, dress, groom, perform bowel movements and urination, go to the toilet, move from the bed to the chair, walk and climb stair. The total score ranges from 0 to 100, with higher scores indicating greater independence (best), and lower scores indicating higher levels of dependence in basic daily activities.
Accelerometer-based physical activity | T0 (baseline) and T1 (post 12 weeks)
  Measurement of physical activity levels (i.e., time spent in light-intensity and moderate-to-vigorous intensity) by accelerometer 24 hours a day for seven consecutive days using a GENEActiv device worn on the non-dominant wrist.
Falls | T0 (baseline) and T1 (post 12 weeks)
  The number of falls in the last year was registered.
Heart rate variability indices from electrocardiogram (ECG) | T0 (baseline) and T1 (post 12 weeks)
  Heart rate variability indices were derived from 10-minute resting recordings using a 12-lead Holter ECG. Both linear indices (time and frequency domains) and non-linear indices (detrended fluctuation ) were calculated from the ECG recording.
Blood pressure | T0 (baseline) and T1 (post 12 weeks)
  Blood pressure is measured in millimeters of mercury (mmHg), including systolic, diastolic, and mean arterial pressure (calculated as diastolic pressure plus one-third of the difference between systolic and diastolic pressures).
Ankle-brachial index relate to blood pressure | T0 (baseline) and T1 (post 12 weeks)
  The ankle-brachial index (ABI) is calculated by measuring systolic pressure in both ankles and both arms. The highest systolic pressure from the arms is used as a reference. The highest systolic pressure from each ankle is divided by this reference to obtain an ABI for each leg. The final ABI value is the lower of the two leg measurements.
Albumin | T0 (baseline) and T1 (post 12 weeks)
  Albumin concentration is measured in blood samples.
C-reactive protein | T0 (baseline) and T1 (post 12 weeks)
  C-reactive protein concentration is measured in blood samples.
inflammatory cytokines | T0 (baseline) and T1 (post 12 weeks)
  Inflammatory cytokines (IL-6 and IL-1β) are measured in blood samples.
Circulating microRNA levels | T0 (baseline) and T1 (post 12 weeks)
  MicroRNAs associated with frailty (miR-194-5p, miR-125b-5p) are measured in blood samples.
Gene expressions of aging (ABLIM1, CCR7, LEF1, EGR1) | T0 (baseline) and T1 (post 12 weeks)
  Gene expressions of aging (ABLIM1, CCR7, LEF1, EGR1) are measured in blood samples.

SECONDARY OUTCOMES:
Resilience | Only baseline (T0)
  The Brief Resilience Scale consists of 6 items designed to measure the ability to recover or "bounce back" from stress. The average score ranges from 1 to 5, and higher values indicate better resilience.

CONTACTS AND LOCATIONS:
Overall Officials: Nuria Garatachea, PhD, Principal Investigator — Universidad de Zaragoza
Locations (1):
- University of Zaragoza, Zaragoza, Zaragoza, Spain